CLINICAL TRIAL: NCT04800614
Title: An Open-label, Randomized, Three-period, Crossover Study of the Effect of Food on the Pharmacokinetics of a Single Oral Dose of Sitravatinib in Healthy Adult Subjects
Brief Title: A Study to Explore the Effect of Food Before a Single Dose of Sitravatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 516-009
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Healthy Adults
MeSH Terms: interventions — sitravatinib

STUDY DESIGN:
Intervention Model Description: Three Period Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Fasted dosing followed by fed dosing (high-fat meal) followed by fed dosing (low-fat meal) (Experimental): Dosing in the fasted state followed by fed dosing after high and low fat meals
  Interventions: Drug: sitravatinib
- Fasted dosing followed by fed dosing (low-fat meal) followed by fed dosing (high-fat meal) (Experimental): Dosing in the fasted state followed by fed dosing after low and high fat meals
  Interventions: Drug: sitravatinib
- Fed dosing (high-fat meal) followed by fasted dosing followed by fed dosing (low-fat meal) (Experimental): Dosing after a high-fat meal followed by doing in the fasted sate followed by dosing after a low-fat meal
  Interventions: Drug: sitravatinib
- Fed dosing (high-fat) followed by fed dosing (low-fat) followed by dosing in the fasted state (Experimental): Fed dosing (high-fate meal) followed by fed dosing (low-fate meal) followed by dosing in the fasted state
  Interventions: Drug: sitravatinib
- Fed dosing (low-fat) followed dosing in the fasted state followed by fed dosing (high fat) (Experimental): Fed dosing (low-fat) meal followed dosing in the fasted state followed by fed dosing (high-fat meal)
  Interventions: Drug: sitravatinib
- Fed dosing (low-fat) followed by fed dosing (high-fat) followed by dosing in the fasted state (Experimental): Fed dosing after a low-fat and high-fate meals followed by dosing in the fasted state
  Interventions: Drug: sitravatinib

INTERVENTIONS:
Drug: sitravatinib — 100 mg sitravatinib on Day 1 of each of 3 periods

SUMMARY:
An Open-label, Randomized, Three-period, Crossover Study of the Effect of Food on the Pharmacokinetics of a Single Oral Dose of Sitravatinib in Healthy Adult Subjects

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at screening and/or check-in
* Females of childbearing potential will not be pregnant or lactating and must have a negative result on an approved pregnancy test at screening and check-in. Females of childbearing potential must agree to use contraception
* Male subjects must agree to use contraception
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions

Key Exclusion Criteria:

* History of drug/chemical abuse within 2 years prior to screening.
* History of alcohol abuse within 12 months prior to screening
* Positive urine drug screen at screening or check-in or positive alcohol test at check-in.
* Use of tobacco- or nicotine-containing products or e-cigarettes (with or without nicotine) within 3 months prior to check-in for Period 1; or positive cotinine at screening or check-in.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days prior to study drug administration on Day 1 of Period 1.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to study drug administration on Day 1 of Period 1.
* Use or intend to use any prescription medications/products within 14 days prior to study drug administration on Day 1 of Period 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax (sitravatinib) | Up to 72 hours after dosing
  Maximum observed plasma concentration
Pharmacokinetics - AUC∞ (sitravatinib) | Up to 72 hours after dosing
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - AUClast (sitravatinib) | Up to 72 hours after dosing
  AUC from time zero to the last measured time point

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to 44 days
  Incidence and severity of adverse events (AEs) dosed in the fasted and fed states in healthy adult subjects

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Chin, MD, Study Director — Mirati Therapeutics
Locations (1):
- Covance Clinical Research Unit, Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No